CLINICAL TRIAL: NCT05234190
Title: A Single-arm, Open-label, Multi-center, Phase I/II Study Evaluating the Safety and Clinical Activity of QEL-001, an Autologous CAR T Regulatory Cell Treatment Targeting HLA-A2, in HLA-A2/ A28neg Patients That Have Received an HLA-A2pos Liver Transplant.
Brief Title: Safety and Clinical Activity of QEL-001 in A2-mismatch Liver Transplant Patients
Acronym: LIBERATE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Quell Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QEL-001-CLN-01; 2021-001379-18 (EudraCT Number)
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Rejection; Transplant, Liver; Liver Failure; Liver Diseases
Keywords: Regulatory T cells; Chimeric Antigen Receptor; Autologous; Genetically modified cells
MeSH Terms: conditions — Rejection, Psychology; Liver Failure; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: QEL-001

INTERVENTIONS:
Drug: QEL-001 — QEL-001 is an autologous therapy that is composed of engineered regulatory T cells transduced with a lentiviral vector containing a CAR directed against HLA-A2. Treatment will be given via an IV infusion.
  Other Names: HLA-A2 CAR-Treg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of QEL-001 in the prevention of liver transplant rejection following immunosuppression withdrawal. QEL-001 is a product made from a patients own cells, which are genetically modified and designed to help the transplant recipient's body accept their donated liver and prevent their immune system from rejecting it once immune suppression is withdrawn.

DETAILED DESCRIPTION:
This study is a multicenter, first-in-human, open-label, single-arm study of an autologous CAR T regulatory (CAR-Treg) in HLA-A2 mismatched liver transplant recipients. The aim is for the CAR-Tregs to be activated on recognition of HLA-A2 antigens present on the donated liver and subsequently induce and maintain immunological tolerance to the organ.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Subject who are HLA A2/A28 negative who have received HLA A2-mismatch liver transplant 12 months to 5 years prior to study entry.
* Able and willing to use contraception.
* Be on stable maintenance of immunosuppression for at least 12 weeks prior to study entry.

Exclusion Criteria:

* Severe cardiac, respiratory disease or any other major organ dysfunction.
* Subjects with prior non-liver solid organ or hematopoietic stem cell transplant.
* Known hypersensitivity to study medication ingredients, protocol defined immunosuppressive medications, or a significant allergic reaction to any drug.
* Positive serology for human immunodeficiency virus (HIV), active or latent tuberculosis (TB) or other clinically active local or systemic infection.
* Use of investigational agents within 3 months of screening.
* Subjects with history of autoimmune disease requiring use of immunosuppression or biologics within 24 months prior to study entry.
* Subject with history of malignancy in the past 5 years.
* Medical or social condition that is not compatible with adequate study follow-up and any other reason that, in the opinion of the Site Investigator or Medical Monitor, would render the subject unsuitable for participation in the study.
* Protocol defined laboratory value for the following parameters:

  * Alanine aminotransferase (ALT) and either alkaline phosphatase (ALP) or gamma-glutamyl transferase (GGT),
  * Kidney function e.g. eGFR,
  * White blood cells,
  * Hemoglobin,
  * Platelets.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2040-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 28 Days post infusion
  Incidence of protocol defined Dose Limiting Toxicities (DLTs).
Long-term safety | Day of infusion through to Week 82 and up to 15 years post infusion
  Incidence and grade of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs) according to CTCAE V5.0.

SECONDARY OUTCOMES:
Immunosuppression related outcome | 2 months and 1 year post withdrawal of immune suppression
  Ability to withdraw immunosuppression (IS) as measured by the percentage of subjects who have stable Liver Function Tests and are IS free at two months and at one year following IS withdrawal.
Tolerance related outcome | 1 year following immune suppression withdrawal
  Ability to achieve operational tolerance as measured by the proportion of subjects meeting the clinical, biochemical and histological operational tolerance criteria at one year following IS withdrawal.
Composite efficacy failure outcome | 1 year following immune suppression withdrawal
  Proportion of subjects with composite event: acute rejection (AR), biopsy proven acute rejection (BPAR), reintroduction of IS or graft loss.

OTHER OUTCOMES:
Assess Safety Related Events | Up to 82 weeks post infusion
  Incidence and severity of infections from treatment to Week 82.
Presence of Replication Competent Lentivirus | up to 52 weeks post infusion
  Absence or presence of exposure to replication-competent lentivirus

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (3):
  - H. Saint Luc, Brussels
  - Hopital Erasme, Brussels
  - UZ Leuven, Leuven
- Spain (3):
  - H. Clinic Barcelona, Barcelona
  - Hospital Reina Sofia, Córdoba
  - G. Gergorio Maranon, Madrid
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No